CLINICAL TRIAL: NCT06954246
Title: A Phase 3, Multicenter, Randomized, Open-label Study of MHB088C for Injection Versus Treatment of Physician's Choice (TPC) in Comparing the Efficacy and Safety in Subjects With Relapsed Small Cell Lung Cancer (SCLC)
Brief Title: A Study of MHB088C Injection Versus Treatment of Physician's Choice in Subjects With Relapsed Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MHB088C-P-301
Record Dates: First submitted 2025-04-18; First posted 2025-05-01 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-04

CONDITIONS: Small Cell Lung Cancer Extensive Stage
Keywords: MHB088C; B7H3; Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Injections; Topotecan; Irinotecan; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MHB088C for Injection (Experimental): Participants randomized to receive 2 mg/kg MHB088C monotherapy on Day 1 and Day 15 of each 28-day cycle until unacceptable toxicity, progressive disease (PD), or withdrawal of consent as specified in the protocol.
  Interventions: Drug: MHB088C for Injection
- Treatment of Physician's Chioce (TPC) (Active Comparator): Participants randomized to receive topotecan, irinotecan, or paclitaxel, as per investigator's choice and per approved label (indicated dose and frequency), until a treatment discontinuation criterion is met as specified in the protocol.
  Interventions: Drug: Topotecan; Drug: Irinotecan; Drug: Paclitaxel

INTERVENTIONS:
Drug: MHB088C for Injection — 2 mg/kg intravenous dose on Day 1 and Day 15 of each 28-day cycle
  Arms: MHB088C for Injection
Drug: Topotecan — 1.25 mg/m^2 intravenous dose on Day 1 to Day 5 of each 21-day cycle
  Arms: Treatment of Physician's Chioce (TPC)
Drug: Irinotecan — 65 mg/m^2 intravenous dose on Day 1 and Day 8 of each 21-day cycle
  Arms: Treatment of Physician's Chioce (TPC)
Drug: Paclitaxel — 135 mg/m^2 intravenous dose on Day 1 of each 21-day cycle
  Arms: Treatment of Physician's Chioce (TPC)

SUMMARY:
This study was designed to compare the efficacy and safety of MHB088C for Injection with treatment of physician's choice (TPC) in participants with relapsed small cell lung cancer (SCLC).

DETAILED DESCRIPTION:
The primary objective of this study is to assess whether treatment with MHB088C for Injection improves prolongs overall survival (OS) compared with treatment of physician's choice among participants with relapsed SCLC.

The secondary objectives of the study are to further evaluate the efficacy/safety of MHB088C for Injection, immunogenicity of MHB088C, and characterize the pharmacokinetics of MHB088C.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all the following criteria to be eligible for randomization into the study:

1. Voluntarily consent to participate in this study and sign the informed consent form.
2. Adults ≥18 years, regardless of gender.
3. ECOG performance status score of 0-1.
4. Estimated survival time of more than 3 months.
5. Capable of understanding trial requirements, willing and able to comply with trial and follow-up procedures.
6. Has histologically or cytologically documented small cell lung cancer (SCLC).
7. Extensive-stage SCLC with disease progression after at least two cycles of platinum-based and PD-1/L1 systemic therapy, with no more than two prior lines of therapy. Prior PD-1/L1 systemic therapy was allowed to use with or without platinum-based regimens.
8. Agrees to provide pre-treatment tumor tissue samples for retrospective analysis of B7-H3 expression and other biomarkers.
9. Has at least 1 measurable lesion according to RECIST v1.1 as assessed by the investigator.
10. Sufficient bone marrow and organ function.

Exclusion Criteria:

Participants who meet any of the following criteria will be disqualified from entering the study:

1. Diagnosis of other primary malignancies within 5 years prior to signing the informed consent form.
2. Prior pathological diagnosis of combined SCLC, or any transformed non-small cell lung cancer or transformed SCLC.
3. Receipt of chemotherapy within 4 weeks prior to the first administration of study drug, or receipt of radiotherapy, biologics, endocrine therapy, immunotherapy, or other anti-tumor therapy within 4 weeks prior to the first dose.
4. Previous or ongoing treatment with topoisomerase I inhibitors, including antibody-drug conjugates (ADCs) containing topoisomerase I inhibitor payloads.
5. Brain metastases (unless asymptomatic and stable for more than 4 weeks prior to randomization); presence of leptomeningeal metastases or brainstem metastases; spinal cord compression (identified via imaging, regardless of symptoms).
6. Bone marrow metastasis.
7. Prior B7-H3-targeted therapy.
8. Has uncontrolled or significant cardiovascular disease.
9. Moderate-to-severe pulmonary disease significantly impairing lung function, including idiopathic pulmonary fibrosis, autoimmune/connective tissue disorders with lung involvement, or prior pneumonectomy.
10. Has history of (non-infectious) interstitial lung disease (ILD)/pneumonitis that required corticosteroids, current ILD/pneumonitis, or suspected ILD/pneumonitis that cannot be ruled out by imaging at Screening.
11. Moderate or severe pulmonary diseases severely affecting lung function.
12. Active tuberculosis, autoimmune diseases not in clinical remission, other acquired or congenital immunodeficiency diseases, or history of allogeneic stem cell, bone marrow, or organ transplantation.
13. Serious infections within 4 weeks before the first dose, including but not limited to those requiring systemic antibiotic therapy, bacteremia, or severe pneumonia.
14. Clinically uncontrolled third-space effusion requiring intervention, including pleural or peritoneal effusions.
15. Known hypersensitivity to investigational product components, analogues, or control drugs (e.g., topotecan, irinotecan, paclitaxel).
16. Pregnant or lactating women, or women/men intending to conceive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | From the date of randomization to the date of death due to any cause, up to approximately 5 years

SECONDARY OUTCOMES:
Number of Participants With Objective Response Rate Assessed by Investigator | Baseline up until documented progressive disease, death, lost to follow-up, or withdrawal by the participant, up to approximately 5 years
  Confirmed objective response rate (ORR) is defined as the sum of the complete response (CR) rate and partial response (PR) rate based on investigator by Response Evaluation Criteria In Solid Tumors (RECIST) v1.1.
Progression-free Survival As Assessed by Investigator | Baseline up until documented progressive disease, death, lost to follow-up, or withdrawal by the participant, up to approximately 5 years
  PFS is defined as the time interval from the date of randomization to the date of disease progression as per investigator assessment or death due to any cause.
Duration of Response As Assessed by Investigator | From the date of first documentation of confirmed response (CR or PR) to the first documentation of objective progression or to death due to any cause, whichever occurs first, up to approximately 5 years
  Duration of response (DoR) is defined as the time from the date of the first documentation of objective response (complete response [CR] or partial response [PR]) to the date of the first documentation of progressive disease (PD) or death. The DoR will be calculated for responding participants (PR or CR) only.
Disease Control Rate As Assessed by Investigator | Baseline up until documented progressive disease, death, lost to follow-up, or withdrawal by the participant, up to approximately 5 years
  Disease control rate is defined as the proportion of participants who have achieved a best overall response of confirmed CR, confirmed PR, or SD (or non-CR/non-PD) by investigator assessment per RECIST v1.1.
Incidence and severity of adverse events (AEs), serious adverse events (SAEs), AEs leading to treatment interruption, and AEs leading to treatment discontinuation. | Baseline up to 5 years
  Assessed based on NCI CTCAE v5.0
Pharmacokinetic Parameter Maximum Concentration for MHB088C, Total Anti-B7-H3 Antibody, and MH30010008 | Day 1 and 15 of Cycle 1 before infusion (BI), end of infusion (EOI), and 5 hours after completion of infusion; Day 1 of Cycle 2 to Cycle 5, BI and EOI; Day 1 of Cycle 6 and every 3 cycles thereafter up to 5 years and EOT visit, BI (each cycle is 28 days)
  Maximum concentration (Cmax) will be assessed using non-compartmental methods in participants randomized to the MHB088C group.
Pharmacokinetic Parameter Time to Maximum Concentration for MHB088C, Total Anti-B7-H3 Antibody, and MH30010008 | Day 1 and 15 of Cycle 1 before infusion (BI), end of infusion (EOI), and 5 hours after completion of infusion; Day 1 of Cycle 2 to Cycle 5, BI and EOI; Day 1 of Cycle 6 and every 3 cycles thereafter up to 5 years and EOT visit, BI (each cycle is 28 days)
  Pharmacokinetic Parameter Time to Maximum Concentration for MHB088C, Total Anti-B7-H3 Antibody, and MH30010008.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, China